CLINICAL TRIAL: NCT07382986
Title: Integrative Medicine Program for COPD With Comorbidity Management
Brief Title: IMPACT COPD Cohort (China)
Acronym: IMPACT
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BeijingCYH-2025ZD0548901
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Multimorbidities
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Real-World Integrative COPD Care and Continuous Multisensor Monitoring — Participants will receive routine clinical care according to GOLD guideline and local clinical practice. This observational cohort collects longitudinal data through conventional clinical assessments (questionnaires, spirometry, imaging, and biomarkers) and continuous multisensor digital monitoring (e.g., heart rate, blood pressure, activity, and sleep), along with digital Traditional Chinese Medicine (TCM) phenotyping (tongue, pulse, and facial features). No study-mandated therapeutic intervention is assigned.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a major chronic respiratory condition with high prevalence of multimorbidity. COPD and comorbidities interact dynamically, contributing to symptom fluctuation, acute exacerbations, hospitalization, and long-term disease progression.

The IMPACT COPD Cohort (China) is a multicenter prospective observational cohort designed to establish a real-world evidence base for integrative Chinese-Western medicine management of COPD with comorbidities. The cohort integrates conventional clinical assessments (symptoms, questionnaires, spirometry, imaging, and biomarkers) with continuous multisensor digital monitoring (e.g., heart rate, blood pressure, activity, sleep patterns, and other physiological and behavioral measures) and digital Traditional Chinese Medicine (TCM) phenotyping (e.g., tongue, pulse, and facial diagnostics).

The study aims to characterize risk profiles of high-risk populations and patients with confirmed comorbidities, develop and validate prediction models for comorbidity risk and acute exacerbation events, and support evidence generation for long-term management strategies with early screening and risk warning capabilities across hospital, community, and home settings.

ELIGIBILITY:
Inclusion Criteria:

Age 40-80 years; Diagnosis of chronic obstructive pulmonary disease (COPD) according to the 2025 GOLD criteria.

Exclusion Criteria:

Acute exacerbation of COPD within the past 4 weeks; Presence of other pulmonary diseases causing chronic respiratory failure in addition to COPD, such as severe bronchiectasis, pneumoconiosis, post-tuberculosis destroyed lung, chest wall deformity, or neuromuscular disease; Cystic fibrosis or interstitial lung disease; Severe respiratory failure requiring long-term mechanical ventilation via tracheostomy; History of lung or other organ transplantation; Severe pleural disease or chest wall abnormalities that interfere with imaging or pulmonary function assessment; Lung cancer or other malignancy with widespread metastatic disease; Previous or current chemotherapy and/or radiotherapy that may affect pulmonary function or structural assessment; Uncontrolled rheumatic/autoimmune diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus); HIV infection; Long-term use of immunosuppressive agents or systemic corticosteroids; Severe organ dysfunction, such as severe cardiac, hepatic, or renal failure, or severe pulmonary arterial hypertension; Hospitalization due to myocardial infarction, heart failure, or other cardiovascular events within the past 3 months; Major surgery involving the chest, abdomen, or eyes within the past 3 months; Presence of intrathoracic metallic foreign bodies or implants that interfere with imaging assessment (e.g., pacemaker, implantable cardioverter-defibrillator, metallic prosthetic valves, other metallic devices, or shrapnel); Allergy to any component of the investigational Chinese herbal compound formula(s); Allergy to any component of ICS+LABA+LAMA therapy or to inhaler propellants/excipients; Unable to accept and wear wearable devices; Pregnant or breastfeeding women; Long-term bedridden status, loss of ability to perform activities of daily living, or life expectancy <1 year; Dementia or other cognitive impairment preventing informed consent and follow-up; Living far from the study center, or planned relocation within the next 3 years, making follow-up infeasible; Current participation in another interventional clinical trial involving the respiratory system; Refusal to provide written informed consent.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from multiple hospitals in China. Eligible participants are adults aged 40-80 years with COPD diagnosed according to the 2025 GOLD criteria, identified in outpatient clinics and/or inpatient settings and enrolled for prospective follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Annual rate of COPD exacerbation | up to 36 months
Incidence of COPD-related comorbidities (hypertension, coronary artery disease, arrhythmia, heart failure, diabetes, etc.) | up to 36 months

IPD SHARING:
Plan to Share IPD: No